CLINICAL TRIAL: NCT00550134
Title: Cognitive Changes Associated With Breast Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); The City College of New York (Other); Brigham and Women's Hospital (Other); Biomedical Engineering Newark College of Engineering New Jersey Institute of Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 07-130
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer; Cognitive Side Effects of Cancer Treatments; Stage I, II and III A Breast Cancer
Keywords: Breast Cancer; Quality of life
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Magnetic Resonance Spectroscopy; Comet Assay; Cellular Senescence; Memory and Learning Tests; Neuropsychological Tests; 2-cyclohexylidenhydrazo-4-phenyl-thiazole; Multicenter Studies as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood

GROUPS / COHORTS (3):
- 1, Non Cancer group: A noncancer control group (N=35), frequency matched on age (< 50 and ≥ 50) and education (less than college or some college and above) will also be recruited and evaluated with the same neuropsychological test battery on a schedule that matches the inter-test interval of the patients.
  Interventions: Behavioral: Questionnaires, MRI, Comet assay and Cell senescence
- 2 Breast Cancer Patients Scheduled for chemotherapy: We will recruit patients with localized breast cancer undergoing adjuvant chemotherapy for the first time and will test the effects of chemotherapy will be given a battery of neuropsychological tests and an MRI evaluation prior to beginning chemotherapy and approximately one month (plus/minus 4 weeks) following completion of treatment.
  Interventions: Behavioral: Questionnaires, MRI, Comet assay and Cell senescence
- 3 Breast Cancer Patients Not Scheduled for Chemotherapy: We will recruit patients with localized breast cancer not undergoing adjuvant chemotherapy.
  Interventions: Behavioral: Questionnaires, MRI, Comet assay and Cell senescence

INTERVENTIONS:
Behavioral: Questionnaires, MRI, Comet assay and Cell senescence — Neuropsychological and psychological testing MRI, Comet assay and Cell senescence
  Other Names: Wide Range Achievement Test - Reading subtest (WRAT 4, 43); Phonemic Verbal Fluency (44); California Verbal Learning Test II (45); Logical Memory I and II (WMS III, 46); Brown Location Test (47); Paced Auditory Serial Addition Test (PASAT, 48); Trail Making Tests (49); The Trail Making Test (Part B); Grooved Pegboard (50); Digit Symbol (WAIS-III, 62); Continuous Performance Test (CPT, 51); Center for Epidemiological Study - Depression (CES-D, 52); Spielberger State Anxiety Inventory (STAI, 53); Fatigue Symptom Inventory (FSI, 54); Functional Assessment of Cancer Therapy-Cognition (FACT-Cog, 55)
  Groups: 1, Non Cancer group
Behavioral: Questionnaires, MRI, Comet assay and Cell senescence — Neuropsychological and psychological testing MRI, Comet assay and Cell senescence
  Other Names: Wide Range Achievement Test -Reading subtest (WRAT 4, 43); Phonemic Verbal Fluency (44); California Verbal Learning Test II (45); Logical Memory I and II (WMS III, 46); Brown Location Test (47); Paced Auditory Serial Addition Test (PASAT, 48); Trail Making Tests (49); The Trail Making Test (Part B); Grooved Pegboard (50); Digit Symbol (WAIS-III, 62); Continuous Performance Test (CPT, 51); Center for Epidemiological Study - Depression (CES-D, 52); Spielberger State Anxiety Inventory (STAI, 53); Fatigue Symptom Inventory (FSI, 54); Functional Assessment of Cancer Therapy-Cognition (FACT-Cog, 55)
  Groups: 2 Breast Cancer Patients Scheduled for chemotherapy
Behavioral: Questionnaires, MRI, Comet assay and Cell senescence — Neuropsychological and psychological testing, MRI, Comet assay and Cell senescence
  Other Names: Wide Range Achievement Test -Reading subtest (WRAT 4, 43); Phonemic Verbal Fluency (44); California Verbal Learning Test II (45); Logical Memory I and II (WMS III, 46); Brown Location Test (47); Paced Auditory Serial Addition Test (PASAT, 48); Trail Making Tests (49); The Trail Making Test (Part B); Grooved Pegboard (50); Digit Symbol (WAIS-III, 62); Continuous Performance Test (CPT, 51); Center for Epidemiological Study - Depression (CES-D, 52); Spielberger State Anxiety Inventory (STAI, 53); Fatigue Symptom Inventory (FSI, 54); Functional Assessment of Cancer Therapy-Cognition (FACT-Cog, 55)
  Groups: 3 Breast Cancer Patients Not Scheduled for Chemotherapy

SUMMARY:
Patients with cancer often complain that their "mind does not seem to be clear." This can be due to stress, depression, anxiety, or physical problems caused by cancer or the treatments used to control symptoms. There are many purposes for this study; one of them is to learn about the effects of cancer treatments on the brain, and another is to identify useful tools to detect these effects. The results of this study may stimulate new research comparing different treatments to the current treatment so the researchers may learn how to treat symptoms more effectively and improve patient quality of life. We would also like to learn more about the effects chemotherapy may have on DNA.

DETAILED DESCRIPTION:
This is a prospective, longitudinal study to examine time-dependent neurocognitive changes in patients with breast cancer receiving adjuvant chemotherapy. This study will assess chemotherapy-induced cognitive dysfunction. The researchers will recruit patients with localized breast cancer undergoing adjuvant chemotherapy for the first time and will test the effects of chemotherapy on patients' cognitive function utilizing a standardized neuropsychological battery. Patients scheduled for chemotherapy will be given a battery of neuropsychological undergo MRI evaluation prior to beginning chemotherapy and one month following completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age but not older than 70years of age
* Patient is female
* Patient is able to understand English, through verbal and written communication
* In the judgment of the investigator and/or the consenting professional patient is able to provide informed consent
* Patient has a diagnosis of breast cancer (stage 0, I, II or IIIA-C), limited to localized disease,
* Patient is chemotherapy naïve and is receiving chemotherapy or is scheduled to receive no chemotherapy as part of adjuvant treatment
* Patient does not report history of prior breast or other cancer with the exception of non-melanoma skin cancer and/or participants who completed treatment for a previous cancer at least 5 years ago and have not undergone any chemotherapy.
* Patient is able to undergo MRI scanning (verified with pre MRI Safety Screening form),
* Patient can comfortably fit inside the MRI machine, verified by back to chest measurement no more than 10 inches or bust circumference of no more than 48 inches.

Exclusion Criteria:

* Patient has documented evidence of cognitive compromise (Blessed- Orientation Memory Cognition Test score > 11
* Patient has a history of neurological disorder with cognitive symptoms (e.g., Alzheimer's disease, Parkinson's disease, multiple sclerosis)
* Patient is Pregnant as confirmed by urine pregnancy test. Participants who are post menopausal or have had a hysterectomy do not need a pregnancy test
* Patient is currently on daily medication for migraine or, insulin-dependent diabetes requiring administration by injection,
* Patient has uncontrollable hypertension as per self report or as documented in the medical record
* Patient has a reported fear of enclosed spaces (Claustrophobia)
* Patient has any of the following items that preclude fMRI evaluation
* Cardiac pacemaker, Joint replacements, Aneurysm clips, Transdermal patched, Aortic clips, Prosthesis, Intracranial bypass clips, Harrington rod , Coronary Artery bypass clips, Biostimulator, Renal Transplant Clips, Bone or joint pins, Other vascular clips or filters, Tissue expander ,Implanted neurostimulators, Metal mesh, Artificial heart valve, Stents, Insulin pump, Wire structures, Electrodes, Shrapnel/bullets, Hearing Aids implant, Implanted electrical devices, IUD, Metal in eyes, Shunts, Ocular Implants, Hair extensions, Hair implants, Tattoos above the waist, Any possible metal in body
* Patient has dentures, body jewelry or wig that they are unable to remove
* History of head injury with evidence of brain injury or loss of consciousness for > 60 minutes or cognitive sequelae
* Untreated or current episode of depression (answering positively to either of the two screening questions from the PHQ-9 (Kroenke, et al., 2001)
* Self-reported sleep disorders that could influence cognitive functioning including sleep apnea and and narcolepsy
* History of Axis I psychiatric disorder (DSM-IV), major affective disorder (untreated), bipolar disorder, schizophrenia disorder (DSM-IV) or substance use disorders (self reported and/or stated in medical record)
* History of schizophrenia, bipolar disorder or substance use disorders
* Patient is unwilling to undergo fMRI component if selected
* Patient has undergone previous chemotherapy treatment

Healthy Control Inclusion Criteria:

* Participant is 18 years of age but not older than 70 years of age,
* Participant is female
* Participant is able to understand English, through verbal and written communication
* In the judgment of the investigator and/or the consenting professional participant is able to provide informed consent
* Patient is able to undergo MRI scanning (verified with pre MRI Safety Screening form)
* Patient can comfortably fit inside the MRI machine, verified by back to chest measurement no more than 10 inches or bust circumference of no more than 48 inches.

Healthy Control Exclusion Criteria:

-Participant has Documented evidence of severe cognitive compromise (Blessed- Orientation Memory Cognition Test score > 11

* Participant has a history of neurological disorder with cognitive symptoms (e.g., Alzheimer's disease, Parkinson's disease, multiple sclerosis).
* Participant is pregnant as indicated by urine pregnancy test,
* As per self report participant is currently on daily medication for migraine, or , insulin dependent diabetes requiring administration by injection,
* As per self report participant has uncontrollable hypertension,
* As per self report, participant has a reported fear of enclosed spaces (Claustrophobia)
* As per self report, participant has any of the following items that preclude fMRI evaluation Cardiac pacemaker, Joint replacements, Aneurysm clips, Transdermal patched, Aortic clips Prosthesis, Intracranial bypass clips, Harrington rod , Coronary Artery bypass clips, Biostimulator, Renal Transplant Clips, Bone or joint pins, Other vascular clips or filters, Tissue expander ,Implanted neurostimulators, Metal mesh, Artificial heart valve, Stents, Insulin pump, Wire structures, Electrodes, Shrapnel/bullets, Hearing Aids implant, Implanted electrical devices, IUD, Metal in eyes, Shunts, Ocular Implants, Hair extensions, Hair implants, Tattoos above the waist, Any possible metal in body
* As per self report, participant has dentures, body jewelry or wig that they are unable to remove
* As per self report, participant has a history of head injury with evidence of brain injury or loss of consciousness for > 60 minutes or cognitive sequelae
* As per self report, participant has untreated or current episode of depression (answering positively to either of the two screening questions from the PHQ-9 (Kroenke, et al., 2001)
* As per self report, participant has sleep disorders that could influence cognitive functioning including sleep apnea and narcolepsy,
* As per self report, participant has history of Axis I psychiatric disorder (DSM-IV), major affective disorder (untreated), bipolar disorder, schizophrenia disorder (DSM-IV) or substance use disorders
* As per self report, participant has undergone previous chemotherapy treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential subjects for the study will be identified MSKCC's clinic.
  Healthy control group participants will be recruited through advertisements and flyers which will be available/advertised in the community. Health control participants will also be recruited by asking survivors if they have a friend who might want to volunteer for the study.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2007-10-24 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
To evaluate changes in cognitive performance pre- to post-chemotherapy in breast cancer patients. | approximately 4 to 6 months from baseline, depending on chemotherapy regimen

SECONDARY OUTCOMES:
To evaluate associations between changes in frontal cortex and hippocampal volumes and activation patterns and changes in neuropsychological test performance. | 4 to 6 months
To evaluate the relationship between change in level of oxidative DNA damage markers of cell senescence (Telomere attrition) and changes in volume and activation patterns in prefrontal cortex and hippocampus. | 4 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tim Ahles, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org